CLINICAL TRIAL: NCT00658437
Title: A Phase II Multicenter Study to Test Progression-free and Overall Survival of CY-503 in the Treatment of Patients With Unresectable Stage IV Metastatic Melanoma After Antineoplastic Treatment Failure
Brief Title: CY503 for the Treatment of Malignant Melanoma Stage IV After Failure of Prior Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytavis Biopharma GmbH (Industry)
Responsible Party: Cytavis Biopharma GmbH, Industry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CY503C1; EudraCT no. 2007-000427-17
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2009-08

CONDITIONS: Melanoma
Keywords: Melanoma, Stage IV, Phase II
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CY-503 — solution for subcutaneous injection, 350 ng twice weekly

SUMMARY:
The trial is designed as a phase II evaluation of the effect of CY-503 on progression free survival (PFS) in patients with stage IV malignant melanoma after failure of prior therapy. The aim of the study is at least a rate of 25% (PFS >/= 3 months).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable, Stage IV metastatic melanoma
* Failure of prior chemotherapy and / or immunotherapy based regimen
* Measurable disease (based on RECIST criteria)
* Males and females of at least 18 years of age
* Women of reproductive potential (defined as being <1 year post-menopausal) must have a negative pregnancy test within 3 days prior to randomization; and men and women of reproductive potential must agree to practice an effective method of avoiding pregnancy
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1.
* Life expectancy of at least 3 months
* WBC ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, platelet count ≥100,000/mm3
* Bilirubin ≤ 1.5 mg/dL (25.65 μmol/L) (unless due to Gilbert's syndrome in which case the bilirubin should be ≤3.5 mg/dL (59.86 μmol/L)), aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 3 × upper limit of normal (ULN); hepatic alkaline phosphatase ≤ 3.0 × ULN
* LDH ≤ 2.5 upper limit of normal (ULN)
* Serum creatinine ≤ 1.5 mg/dL (132.60 μmol/L), proteinuria < 2.0 g/24 hr urine
* Patients who have had prior treatment with adjuvant or palliative immunotherapy are eligible provided that therapy ended at least 1 month prior to randomization and all treatment-related toxicities have resolved
* Patients with bone metastasis should be evaluated by the investigator and prior treatment should be finished at least 1 month prior to randomization
* Prior radiotherapy (for palliative care only) is allowed provided there is measurable/evaluable disease outside of the radiation field and all radiation-related toxicities have resolved; if there is only one measurable lesion it may not have been irradiated unless subsequent progression has been documented
* Patients who had prior major surgery are eligible if at least 4 weeks have passed since their surgery and all surgical wounds have healed prior to randomization and at least one measurable tumor is present
* All toxicities related to prior adjuvant therapy must have resolved
* Written informed consent

Exclusion Criteria:

* Pregnancy or nursing
* Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for treatment of cancer
* Current or planned participation in a research protocol
* Received an investigational agent within 4 weeks prior to randomization
* Brain metastases or primary brain tumors, symptomatic pleural effusion or ascites requiring paracentesis
* Ocular melanoma
* History of prior malignancies within the past 5 years other than non-melanomatous skin cancers that have been controlled, carcinoma in situ of the cervix, T1a or b prostate cancer noted incidentally during a transurethral resection of prostate (TURP) with prostate-specific antigen (PSA) values within normal limits since TURP, or superficial bladder cancer
* Any evidence of or history elicited by the investigator of symptomatic cerebrovascular events within 6 months prior to randomization; or any history or evidence of pulmonary embolism or thrombophlebitis requiring anticoagulant therapy
* Any current evidence of hematemesis, melena, hematochezia, or gross hematuria
* Elective surgery planned during the study period through 30 days after the last dose of CY-503
* History of hypersensitivity to previously administered mistletoe
* Prior therapy with mistletoe
* History of primary immunodeficiency
* Known human immunodeficiency virus (HIV) or known active viral hepatic infections
* Prior treatment with CY-503
* A general medical or psychological condition or behaviour in the opinion of the investigator, might not permit the patient to complete the study or sign the informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Tumor assessment by CT and MRT | each 8 weeks

SECONDARY OUTCOMES:
Immunological response (e.g. measurement of cytokines in serum) | each 4 weeks
Assessment of quality of life using a standardized questionnaire | each 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mohr, MD, Principal Investigator — Elbe Klinikum Buxtehude, Germany
Locations (4):
- Germany (4):
  - Haut Tumor Zentrum Charité, Berlin
  - Dermatologisches Zentrum Elbe-Klinikum Buxtehude, Buxtehude
  - Hautklinik Linden MH Hannover, Hanover
  - Universitäts-Hautklinik Kiel, Kiel

REFERENCES:
- [Derived] Trefzer U, Gutzmer R, Wilhelm T, Schenck F, Kahler KC, Jacobi V, Witthohn K, Lentzen H, Mohr P. Treatment of unresectable stage IV metastatic melanoma with aviscumine after anti-neoplastic treatment failure: a phase II, multi-centre study. J Immunother Cancer. 2014 Aug 19;2:27. doi: 10.1186/s40425-014-0027-z. eCollection 2014. PMID 25324973